CLINICAL TRIAL: NCT06764771
Title: A Phase 1/1b Open-label Study of BMS-986488 as Monotherapy and Combination Therapy in Participants With Advanced Malignant Tumors
Brief Title: A Study of BMS-986488 as Monotherapy and Combination Therapy in Participants With Advanced Malignant Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA234-0001
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Tumors
Keywords: Colorectal Cancer; CRC; Renal Cell Carcinoma; RCC; Non-Small Cell Lung Cancer; NSCLC; Cancer; Oncology; Phase 1; Solid Tumor
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — adagrasib; Cetuximab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1A: BMS-986488 Monotherapy (Experimental)
  Interventions: Drug: BMS-986488
- Part 1B: BMS-986488 + Adagrasib (Experimental)
  Interventions: Drug: BMS-986488; Drug: Adagrasib
- Part 1C: BMS-986488 + Adagrasib + Cetuximab (Experimental)
  Interventions: Drug: BMS-986488; Drug: Adagrasib; Drug: Cetuximab
- Part 1D: BMS-986488 + Nivolumab (Experimental)
  Interventions: Drug: BMS-986488; Drug: Nivolumab
- Part 2A: BMS-986488 Monotherapy (Experimental)
  Interventions: Drug: BMS-986488
- Part 2B: BMS-986488 + Adagrasib (Experimental)
  Interventions: Drug: BMS-986488; Drug: Adagrasib
- Part 2C: BMS-986488 + Adagrasib + Cetuximab (Experimental)
  Interventions: Drug: BMS-986488; Drug: Adagrasib; Drug: Cetuximab
- Part 2D: BMS-986488 + Nivolumab (Experimental)
  Interventions: Drug: BMS-986488; Drug: Nivolumab

INTERVENTIONS:
Drug: BMS-986488 — Specified dose on specified days
Drug: Adagrasib — Specified dose on specified days
  Other Names: KRAZATI; BMS-986503; MRTX849
  Arms: Part 1B: BMS-986488 + Adagrasib; Part 1C: BMS-986488 + Adagrasib + Cetuximab; Part 2B: BMS-986488 + Adagrasib; Part 2C: BMS-986488 + Adagrasib + Cetuximab
Drug: Cetuximab — Specified dose on specified days
  Other Names: ERBITUX
  Arms: Part 1C: BMS-986488 + Adagrasib + Cetuximab; Part 2C: BMS-986488 + Adagrasib + Cetuximab
Drug: Nivolumab — Specified dose on specified days
  Other Names: OPDIVO; BMS-936558
  Arms: Part 1D: BMS-986488 + Nivolumab; Part 2D: BMS-986488 + Nivolumab

SUMMARY:
This purpose of this study is to determine if experimental treatment with BMS-986488, alone, or in combinations is safe, tolerable, and has anti-cancer activity in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age.
* Histologically confirmed diagnosis of a locally advanced and unresectable or metastatic solid tumor malignancy with any of the following tumor types:.
* Part 1A: clear-cell renal cell carcinoma (ccRCC), clear-cell ovarian cancer (ccOC), non-small cell lung cancer (NSCLC), colorectal cancer (CRC), and pancreatic ductal adenocarcinoma (PDAC).
* Parts 2A, 1D, 2D: ccRCC.

  i) Part 1B: solid tumors with KRAS G12C mutation.

ii) Part 2B: NSCLC with KRAS G12C mutation.

iii) Parts 1C, 2C: colorectal cancer (CRC) with KRAS G12C mutation.

* Participants must have an Eastern Cooperative Oncology Groups (ECOG) Performance Status of 0 or 1.
* Participants must have measurable disease per RECIST v1.1.

Exclusion Criteria:

* Untreated central nervous system (CNS) metastases.
* Leptomeningeal metastasis (carcinomatous meningitis).
* Impaired cardiac function or clinically significant cardiac disease.
* For Parts 1B, 1C, 2B, 2C only (combination with adagrasib):.

  i) History of pneumonitis or interstitial lung disease (ILD).

ii) History of prior severe cutaneous adverse reactions (SCARs), including Stevens-Johnson syndrome (SJS) and toxic epidermal necrolysis (TEN).

- Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Until the end of the Safety Follow-up period (up to approximately 100 days after last dose)
Number of participants with Serious AEs (SAEs) | Until the end of the Safety Follow-up period (up to approximately 100 days after last dose)
Number of participants with AEs meeting protocol-defined Dose-Limiting Toxicity (DLT) criteria | From first dose of study treatment until end of cycle 1 (1 Cycle = 28 Days)
Number of participants with AEs leading to discontinuation | Until the end of the Safety Follow-up period (up to approximately 100 days after last dose)
Number of deaths | From time of informed consent up to 52 weeks after end of treatment visit

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Until Cycle 4, Day 1 (1 Cycle = 28 Days)
Time of maximum observed concentration (Tmax) | Until Cycle 4, Day 1 (1 Cycle = 28 Days)
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Until Cycle 4, Day 1 (1 Cycle = 28 Days)
Objective response rate (ORR) | From time of informed consent up to 52 weeks after end of treatment visit
  Defined as the proportion of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Disease control rate (DCR) | From time of informed consent up to 52 weeks after end of treatment visit
  Defined as the proportion of participants who achieve a best response of CR, PR, or stable disease (SD) assessed by the investigator using RECIST v1.1
Duration of response (DOR) | From time of informed consent up to 52 weeks after end of treatment visit
  Defined as the time between the date of first documented response (CR or PR) to the date of the first documented disease progression as assessed by the investigator using RECIST v1.1 or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (3):
  - Local Institution - 0021, Hackensack, New Jersey
  - Local Institution - 0020, Allentown, Pennsylvania
  - Local Institution - 0024, Germantown, Tennessee
- Local Institution - 0031, Brisbane, Queensland, Australia
- Canada (3):
  - Local Institution - 0032, Vancouver, British Columbia
  - Local Institution - 0015, Montreal, Quebec
  - Local Institution - 0016, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06764771.html